CLINICAL TRIAL: NCT03070990
Title: An Open-label, Randomized, Phase 1 Safety and Pharmacokinetic Study of Enfortumab Vedotin (ASG-22CE) in Japanese Patients With Locally Advanced or Metastatic Urothelial Carcinoma
Brief Title: A Study of Enfortumab Vedotin in Japanese Subjects With Locally Advanced or Metastatic Urothelial Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7465-CL-0101
Record Dates: First submitted 2017-03-01; First posted 2017-03-06 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Urothelial Cancer
Keywords: Urothelial Carcinoma; Enfortumab vedotin; ASG-22CE; Padcev; ASG-22ME; Metastatic Urothelial Cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — enfortumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A: Enfortumab vedotin 1.0 mg/kg (Experimental): All subjects assigned will receive a single 30 minute intravenous infusion of enfortumab vedotin (ASG-22CE) once weekly for 3 weeks of every 4 weeks (i.e., on Days 1, 8, and 15). A cycle is 28 days.
  Interventions: Drug: Enfortumab vedotin
- Arm B: Enfortumab vedotin 1.25 mg/kg (Experimental): All subjects assigned will receive a single 30 minute intravenous infusion of enfortumab vedotin (ASG-22CE) once weekly for 3 weeks of every 4 weeks (i.e., on Days 1, 8, and 15). A cycle is 28 days.
  Interventions: Drug: Enfortumab vedotin

INTERVENTIONS:
Drug: Enfortumab vedotin — All subjects assigned will receive a single 30 minute intravenous infusion of enfortumab vedotin (ASG-22CE) once weekly for 3 weeks of every 4 weeks (i.e., on Days 1, 8, and 15). A cycle is 28 days.
  Other Names: ASG-22CE; Padcev

SUMMARY:
The objective of this study is to assess the safety, tolerability and pharmacokinetics of enfortumab vedotin (ASG-22CE) when administered intravenously to Japanese subjects with locally advanced or metastatic urothelial carcinoma. This study will also assess the immunogenicity as defined by the incidence of anti-drug antibody (ADA) and anti-tumor activity of enfortumab vedotin (ASG-22CE) when administered intravenously to Japanese subjects with locally advanced or metastatic urothelial carcinoma.

DETAILED DESCRIPTION:
All subjects will receive a single 30 minute intravenous (IV) infusion of enfortumab vedotin (ASG-22CE) once weekly for 3 weeks of every 4 weeks (i.e., on Days 1, 8, and 15). A cycle is 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have histologically confirmed, locally advanced (TNM classification T3b and any N; or T and N2-3) or metastatic Transitional Cell Carcinoma of the Urothelium (TCCU) (i.e., cancer of the bladder, renal pelvis, ureter, or urethra). Subjects with Urothelial Carcinoma with squamous differentiation or mixed cell types are eligible.
* Subject must be able to submit a tumor tissue samples for Nectin-4 expression analysis at central laboratory.
* Subject must have failed at least one prior chemotherapy regimen for advanced disease. Urothelial and bladder cancer subjects are not required to have failed prior chemotherapy regimen if considered unfit for cisplatin-based chemotherapy.
* Subject must have measurable disease according to Response Evaluation Criteria in Solid Tumor (RECIST) (version 1.1).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

* Preexisting sensory neuropathy Grade ≥ 2.
* Preexisting motor neuropathy Grade ≥ 2.
* Uncontrolled central nervous system metastasis that requires active treatment.
* Any anticancer therapy within 14 days prior to the first dose of study drug.
* Subjects with pre-existing immunotherapy-related adverse events requiring high doses of systemic steroids are not eligible.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-02-25 (Actual)

PRIMARY OUTCOMES:
Safety assessed by incidence of adverse events | Up to 12 months
  Adverse events will be coded using MedDRA. Adverse events collection begins after signing informed consent and collected until 28 days after the last dose of study drug.
Safety assessed by laboratory tests: Hematology | Up to 12 months
  Descriptive statistics will be used to summarize results.
Safety assessed by laboratory tests: Biochemistry | Up to 12 months
  Descriptive statistics will be used to summarize results.
Safety assessed by laboratory tests: Urinalysis | Up to 12 months
  Descriptive statistics will be used to summarize results.
Safety assessed by laboratory tests: Coagulation studies | Up to 12 months
  Descriptive statistics will be used to summarize results.
Number of participants with vital sign abnormalities and/or adverse events | Up to 12 months
  Number of participants with potentially clinically significant vital sign values.
Safety assessed by electrocardiogram (ECG) | Up to 12 months
  Before measurement of ECGs, the participant should be resting in a supine position for at least 5 minutes. The investigator will assess the ECG charts as "normal", "abnormal (not clinically significant)" or "abnormal (clinically significant)". "Abnormal (not clinically significant)" and "abnormal (clinically significant)" findings will be recorded.
Pharmacokinetics (PK) parameter for total antibody (TAb): Concentration at the end of infusion (CEOI) | Days 1-4, 8, 15-18, 22 of Cycle 1, Day 1 of Cycle 2 and 3, and subsequent cycles up to an average of 12 months
  CEOI will be derived from the PK blood samples collected.
Pharmacokinetics (PK) parameter for antibody drug conjugate (ADC): CEOI | Days 1-4, 8, 15-18, 22 of Cycle 1, Day 1 of Cycle 2 and 3, and subsequent cycles up to an average of 12 months
  CEOI will be derived from the PK blood samples collected.
Pharmacokinetics (PK) parameter for Monomethyl Auristatin E (MMAE): CEOI | Days 1-4, 8, 15-18, 22 of Cycle 1, Day 1 of Cycle 2 and 3, and subsequent cycles up to an average of 12 months
  CEOI will be derived from the PK blood samples collected.
PK parameter for TAb: Maximum observed concentration (Cmax) | Days 1-4, 8, 15-18, 22 of Cycle 1, Day 1 of Cycle 2 and 3, and subsequent cycles up to an average of 12 months
  Cmax will be derived from the PK blood samples collected.
PK parameter for ADC: Cmax | Days 1-4, 8, 15-18, 22 of Cycle 1, Day 1 of Cycle 2 and 3, and subsequent cycles up to an average of 12 months
  Cmax will be derived from the PK blood samples collected.
PK parameter for MMAE: Cmax | Days 1-4, 8, 15-18, 22 of Cycle 1, Day 1 of Cycle 2 and 3, and subsequent cycles up to an average of 12 months
  Cmax will be derived from the PK blood samples collected.
PK parameter for TAb: Trough concentration (Ctrough) | Days 1-4, 8, 15-18, 22 of Cycle 1, Day 1 of Cycle 2 and 3, and subsequent cycles up to an average of 12 months
  Ctrough will be derived from the PK blood samples collected.
PK parameter for ADC: Ctrough | Days 1-4, 8, 15-18, 22 of Cycle 1, Day 1 of Cycle 2 and 3, and subsequent cycles up to an average of 12 months
  Ctrough will be derived from the PK blood samples collected.
PK parameter for MMAE: Ctrough | Days 1-4, 8, 15-18, 22 of Cycle 1, Day 1 of Cycle 2 and 3, and subsequent cycles up to an average of 12 months
  Ctrough will be derived from the PK blood samples collected.
PK parameter for TAb: Time to maximum concentration (Tmax) | Days 1-4, 8, 15-18, 22 of Cycle 1, Day 1 of Cycle 2 and 3, and subsequent cycles up to an average of 12 months
  Tmax will be derived from the PK blood samples collected.
PK parameter for ADC: Tmax | Days 1-4, 8, 15-18, 22 of Cycle 1, Day 1 of Cycle 2 and 3, and subsequent cycles up to an average of 12 months
  Tmax will be derived from the PK blood samples collected.
PK parameter for MMAE: Tmax | Days 1-4, 8, 15-18, 22 of Cycle 1, Day 1 of Cycle 2 and 3, and subsequent cycles up to an average of 12 months
  Tmax will be derived from the PK blood samples collected.
PK parameter for TAb: Partial area under the serum concentration-time curve after first dose and as appropriate (AUC0-7) | Days 1-4, 8, 15-18, 22 of Cycle 1, Day 1 of Cycle 2 and 3, and subsequent cycles up to an average of 12 months
  AUC0-7 will be derived from the PK blood samples collected.
PK parameter for ADC: AUC0-7 | Days 1-4, 8, 15-18, 22 of Cycle 1, Day 1 of Cycle 2 and 3, and subsequent cycles up to an average of 12 months
  AUC0-7 will be derived from the PK blood samples collected.
PK parameter for MMAE: AUC0-7 | Days 1-4, 8, 15-18, 22 of Cycle 1, Day 1 of Cycle 2 and 3, and subsequent cycles up to an average of 12 months
  AUC0-7 will be derived from the PK blood samples collected.
PK parameter for TAb: Terminal or apparent terminal half-life (t1/2) | Days 1-4, 8, 15-18, 22 of Cycle 1, Day 1 of Cycle 2 and 3, and subsequent cycles up to an average of 12 months
  T1/2 will be derived from the PK blood samples collected.
PK parameter for ADC: t1/2 | Days 1-4, 8, 15-18, 22 of Cycle 1, Day 1 of Cycle 2 and 3, and subsequent cycles up to an average of 12 months
  T1/2 will be derived from the PK blood samples collected.
PK parameter for MMAE: t1/2 | Days 1-4, 8, 15-18, 22 of Cycle 1, Day 1 of Cycle 2 and 3, and subsequent cycles up to an average of 12 months
  T1/2 will be derived from the PK blood samples collected.

SECONDARY OUTCOMES:
Incidence of Anti-Drug Antibody (ADA) | Up to 12 months
  Blood samples for anti-drug antibody (ADA) analysis will be collected.
Overall Response Rate | Up to 12 months
  Defined as the proportion of subjects whose best overall response is rated as complete response (CR) or partial response (PR)
Disease Control Rate | Up to 12 months
  Defined as the proportion of subjects whose best overall response is rated as CR, PR, or stable disease (SD)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (8):
- Japan (8):
  - Site JP00003, Tsukuba, Ibaraki
  - Site JP00005, Sendai, Miyagi
  - Site JP00008, Suita, Osaka
  - Site JP00004, Chuo-ku, Tokyo
  - Site JP00007, Koto-ku, Tokyo
  - Site JP00006, Fukuoka
  - Site JP00001, Niigata
  - Site JP00002, Okayama

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Takahashi S, Uemura M, Kimura T, Kawasaki Y, Takamoto A, Yamaguchi A, Melhem-Bertrandt A, Gartner EM, Inoue T, Akazawa R, Kadokura T, Tanikawa T. A phase I study of enfortumab vedotin in Japanese patients with locally advanced or metastatic urothelial carcinoma. Invest New Drugs. 2020 Aug;38(4):1056-1066. doi: 10.1007/s10637-019-00844-x. Epub 2019 Aug 14. PMID 31444589
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/hcp/study.aspx?ID=365